CLINICAL TRIAL: NCT01973803
Title: Clinical Evaluation of the Articulinx InterCarpoMetacarpal Cushion (ICMC) for Osteoarthritis of the First Metacarpal Joint
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Articulinx (Industry)
Responsible Party: Sponsor
Other Study IDs: CL 0030
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Osteoarthritis of the CMC-1 Joint
Keywords: Carpometacarpal joint; Osteoarthritis of CMC-1 joint

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to evaluate the performance of the Articulinx ICMC (InterCarpoMetacarpalCushion) in the carpometacarpal joint (CMC joint) and to describe the clinical results in patients who have been treated with this device. Expected results include the relief of symptoms and improvement of function in patients with symptomatic osteoarthritis (OA) of the CMC-1 joint. Evaluation of device performance will be achieved through measurements of pain, pain medication use, and joint function in up to 40 subjects. Each subject will be compared to their pre-surgery status for each endpoint.

DETAILED DESCRIPTION:
The Articulinx ICMC is intended to be implanted into the basilar, or first carpometacarpal (CMC) joint, as an interpositional spacer between the first metacarpal and trapezium bones. The device is intended to be used in the treatment of thumb disabilities resulting from osteoarthritis of the CMC-1 joint.

The primary objective is to document the performance of the Articulinx ICMC by evaluating pain relief in the CMC joint following device implantation. CMC-1 joint function will be assessed by measurement of lateral key and tripod pinch strength, grip strength, and range of motion. Patient reported physical functioning and symptoms will be measured by DASH scores. Trapezial height will be measured on standard PA xrays of the CMC joint. Incidence of unanticipated device and procedure related adverse events will be documented intraoperatively through one year follow-up.

Primary and secondary outcomes will be evaluated through one year and subjects will continue to be followed for two years for evaluation of longer term performance.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed by the investigator to be medically acceptable for a surgical procedure
* Patient is aged 40 to 75 inclusive
* Patient has symptomatic osteoarthritis of the carpometacarpal (CMC-1) joint as demonstrated by a minimum DASH score of 40 at baseline
* Patient has pain in the target CMC joint as demonstrated by an average VAS pain score greater than or equal to 40 at baseline on a 100mm VAS
* Patient has radiographic evidence of Stage II OA with no free-floating bodies in the CMC-1 joint
* Patient has subluxation of less than one-third of the target CMC joint
* Patient agrees to return to the clinic for follow-up visits at the required times per protocol and follow the requirements of this protocol
* Patient is able and willing to provide voluntary consent to participate

Exclusion Criteria:

* Patient has non-symptomatic osteoarthritis of the first CMC joint
* Patient has small bone or calcific fragments (spurs, osteophytes) in the target CMC joint greater than two millimeters (>2mm) in diameter
* Patient has free floating bodies of any size within the target CMC joint
* Patient has radiographic/imaging evidence of significant osteoarthritic changes within the first metacarpal, or scaphotrapezotrapezoidal (STT) joint of the target wrist consistent with Stage III/IV OA, according to Eaton-Glickel
* Patient has concomitant musculoskeletal pathology of the target hand, such as carpal tunnel syndrome, palmar tenosynovitis, schaphoulnate ligament instability/degeneration, ulnocarpal impaction syndrome, or trigger finger
* Patient has concomitant rheumatic disease (e.g., inflammatory rheumatoid arthritis, cutaneous psoriasis, polyarticular chondrocalcinosis, gout, fibromyalgia) or exhibits signs of metabolic disorders affecting the bone or joint (e.g., osteoporosis,osteomalacia, hyper- or hypo-parathyroidism,Paget's disease)
* Patient has an active infection, sepsis or osteomyelitis
* Patient has skin disease or eruption at the CMC target site
* Patient had previous surgery on the target CMC joint or; prior surgery within the previous 12 months on the wrist of the target hand that could alter the biomechanics of the wrist or CMC-1 joint or; prior surgery on the wrist of the target hand more than 12 months previously fro which there are existing sequelae
* Patient had significant injury to the target CMC joint within the 6 months prior to study enrollment or a significant permanent injury at any time prior to study enrollment
* Patient has a significant comorbid medical condition that could exacerbate pain symptoms or adversely affect physical functioning or healing of the thumb CMC joint (e.g. de Quervains disease, Ehler-Danlos Syndrome, Complex Regional Pain Syndrome)
* Patient has had corticosteroid injections in the target CMC joint within 6 months prior to study enrollment
* Patient takes concomitant immunosuppressive therapy (e.g., oral/injectable glucocorticoids, alkylating agents, antimetabolites, antibodies, drugs acting on immunophilins [Ciclosporin, Sirolimus], interferons, opioids) that could adversely affect healing
* Patient has uncontrolled diabetes mellitus
* Patient takes anticoagulation and or antiplatelet therapy that cannot be stopped prior to surgery
* Patient is planning a pregnancy, or patient is pregnant and/or lactating
* Patient is participating in any other clinical investigation that could impact the outcome of this study
* Patient has a known history of drug or alcohol abuse in the previous 12 months
* Patient has a history of, or is currently engaged in, litigation for musculoskeletal injuries or disorders or medical malpractice
* Patient has other life circumstances that the Investigator feels would interfere with study participation such as planned relocation, difficulty complying with schedule of study follow-up visits, is generally uncooperative

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with early stage carpometacarpal-1 (CMC-1 joint osteoarthritis who may seek treatment at physician hand clinics and community general practitioner clinics.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Average CMC joint pain score | One year
  The post-operative VAS pain score will be compared to pre-operative baseline VAS pain score at one year.

SECONDARY OUTCOMES:
Change in joint function | One year
  Change in joint function post-procedure compared to pre-operative baseline. Measurements of contralateral hand function will be taken at baseline and at subsequent follow-up visits through one year.
Change in DASH scores | One year
  Change in DASH scores post-procedure as compared to pre-operative baseline
Maintenance of trapezial joint space height | One year
  Maintenance of trapezial joint space height compared to pre-operative baseline.
Incidence of unanticipated device and procedure related adverse events | One year
  Incidence of unanticipated device and procedure related adverse events intraoperatively and through one year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Rainer Meffert, MD, Principal Investigator — University of Wurzburg, Klinik und Poliklinik für Unfall-, Hand-, Plastische und Wiederherstellungschirurgie
Locations (3):
- Germany (3):
  - Stiftungsklinikum Mittelrhein, Koblenz
  - Berufsgenossenschaftliche (B-G) Unfallklinik Tübingen, Tübingen
  - University of Wurzburg, Klinik und Poliklinik für Unfall-, Hand-, Plastische und Wiederherstellungschirurgie, Würzburg